CLINICAL TRIAL: NCT06799897
Title: Natural Course of Initially Metabolic Healthy Obese Individuals (Healthy Obesity)?
Status: Recruiting | Type: Observational
Sponsor: ETH Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-03031
Record Dates: First submitted 2024-07-18; First posted 2025-01-29 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy Obesity, Metabolically
Keywords: Obesity; Healthy
MeSH Terms: conditions — Obesity, Metabolically Benign; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main goal of this study is to gain a thorough understanding, which specific factors drive the unhealthy sequelae of obesity. Therefore, the investigators want to understand:

1. What distinguishes obese persons without metabolic diseases from those with medical diseases in a cross-sectional comparison?
2. Which factors drive the conversions from metabolically healthy obesity into a metabolically unhealthy obesity in a longitudinal approach?

DETAILED DESCRIPTION:
The hypothesis is, that changes in the molecular regulation of adipose tissue as well as in adipose tissue cellular composition are responsible for the development of a rather metabolic healthy or unhealthy phenotype. Knowledge of these factors will be used to generate new diagnostic concepts for personalized risk prediction and will furthermore serve as the basis to develop novel strategies to target adipose tissue to improve metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age between 18 and 60 years
* BMI 30-50 kg/m2
* Knowledge of German, which requires sufficient written and allow oral patient education

Inclusion criteria for initially healthy group

* Blood pressure < 140/90 mmHg
* Normal glucose metabolism

  * HbA1c < 6.5 %
  * Fasting Glucose < 7.0 mmol/l
* Normal lipid metabolism

  o LDL-cholesterol < 5.0 mmol/l
* ≤ 2 of the following metabolic syndrome criteria combined (excluding waist circumference)
* TG > 1.7 mmol/l
* HDL-cholesterol > 1.0 mmol/l (male) / > 1.3 mmol/l (female)
* Fasting glucose ≥ 5.6 mmol/l
* BP ≥ 130/85 mmHg

Exclusion Criteria:

* Pregnancy
* Medication and / or pathologies that prevent a safe execution of the fat tissue biopsies
* History of or planned bariatric operation
* Medical conditions that prevent examinations and testing (e.g. symptomatic cardiovascular diseases)
* Active Malignant tumor (<2a remission)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: obese participants
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-01-18 (Estimated); Study Completion 2026-01-18 (Estimated)

PRIMARY OUTCOMES:
Rate of conversion | Conversion will be driven by the occurrence of pathological findings caused by obesity (metabolic or cardiovascular pathologies). Through study completion, an average of 1 year.
  The primary endpoint is the conversion (through study completions, 10 years) from obese but metabolically healthy subjects into obese patients in a pathological metabolic state, through study completion an average of 1 year.

SECONDARY OUTCOMES:
Rate of identification of factors | Conversion will be driven by the occurrence of pathological findings caused by obesity (metabolic or cardiovascular pathologies), through study completion, an average of 1 year.
  The secondary endpoint is the identification of factors alone or in combination (through study completions, 10 years), that related to this conversion from healthy into pathological obesity. This includes factors like: DEXA scans, White Adipose Tissue, lipid and glucose metabolism, vital signs, physical activity, general health and quality of life status...

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Goldhahn, Prof., Study Chair — dTIP / ETH Zürich
Locations (1):
- dTIP / ETH Zürich, Baden, Switzerland